CLINICAL TRIAL: NCT06440785
Title: The Relation Between Following Taylor Swift on Social Media, Connecting With Her Music and Mental Health Outcomes in Youths: Cross-sectional Survey Study
Brief Title: Taylor Swift and Mental Health Outcomes
Status: Recruiting | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: NUS-IRB-2023-864B
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Social Stigma; Psych; Depression, Anxiety; Stress
Keywords: Pop-Culture; Music; Mental Health literacy; Adolescent Health
MeSH Terms: conditions — Social Stigma; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study in Singapore will explore the potential of pop culture, particularly Taylor Swift's music, in influencing young adults' attitudes toward mental health. With the highest prevalence of mental illness among this age group, the study will aim to investigate whether engagement with Swift's songs and social media will be associated with attitudes crucial for help-seeking, such as recognizing mental health issues and being open to professional services. Conducting a survey of over 600 young adults, the researchers will assess participants' mental health symptoms, engagement with Swift's content, social media and demographics, mental health help-seeking attitude and mental health self-diagnosing behavior.

DETAILED DESCRIPTION:
Background: Epidemiological surveys suggest that young adulthood is the age group with the highest prevalence of mental illness. However, many young adults have negative views towards help-seeking and do not access professional services. To address this gap, popular culture may provide population-level levers to improve mental health outcomes.

Objective: In this study, we will focus on Taylor Swift - a singer whose songs explore themes related to mental health. As the first objective, we will seek to understand whether young adults will feel a personal connection to her mental health-themed songs and follow her on social media. We will then examine whether these forms of engagement will predict attitudes critical for help-seeking: namely, acknowledgement that one may have a mental illness, and willingness to seek professional services as needed.

Methods: In the months leading up to Taylor Swift's concerts, we will conduct a survey of over 600 young adults in Singapore (aged 18 to 34). As the primary outcome measures, participants will complete the Self-Identification as Having Mental Illness Scale (SELFI) and the Inventory of Attitudes toward Seeking Mental Health Services scale (IASMHS). As predictor variables, participants will answer questions related to: (i) their baseline symptoms of depression, anxiety, and stress; (ii) their engagement with Taylor Swift's songs and social media content; and (iii) their demographics.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment is restricted to healthy adults between 18-34
* Use at least one of the following social media platforms: Facebook, Instagram, LinkedIn, X (Twitter), TikTok
* Have lived in Singapore for at least 2 years.
* Participants need to be able to read and understand English.

Exclusion Criteria:

* Anyone who does not feel comfortable answering questions related to mental health and exposure to mental health-related content online.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruiting a representative sample of around 600 people through the National University of Singapore (NUS) and the general public in Singapore through physical posters or online platforms (e.g., the university's Work Scheme website, and research groups on Telegram).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Help-Seeking Behaviors | Through study completion, an average of 1 year
  Inventory of Attitudes toward Seeking Mental Health Services (IASMHS). Items were on a 5-point Likert scale ranging from 0 ("Somewhat Disagree") to 4 ("Agree").
Self-Diagnosing Behaviors for Mental Health | Through study completion, an average of 1 year
  Self-identification as having a Mental Illness (SELF-I) scale. Items were on 5-point Likert scale ranging from 1 (Not true at all) to 5 (Completely True)

CONTACTS AND LOCATIONS:
Overall Officials: Sundarimaa Erdembileg, Principal Investigator — Yale-NUS College
Locations (1):
- Yale-NUS, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Given the sensitivity of mental health disclosures and the age of the population, no individual participant data will be shared as agreed upon with the IRB. Results will be published by the investigators in academic journals. Sharing of generated study data can be made available upon request by writing to the investigator(s).